CLINICAL TRIAL: NCT01199549
Title: Phase 1 Bioavailability Study of Different Dietary Antioxidants in Volunteers
Brief Title: Bioavailability Study of Different Dietary Antioxidants in Volunteers
Status: Completed | Type: Observational
Sponsor: Cambridge Theranostics Ltd (Industry)
Responsible Party: Medical Director Dr Ivan Petyaev, Cambridge Theranostics Ltd
Other Study IDs: DAO09C01
Record Dates: First submitted 2010-09-07; First posted 2010-09-13 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Lycopene group: Mixed age and gender group of healthy volunteers for testing bio-availability of Lycopene containing supplement
- Resveratrol group: Mixed age and gender group of healthy volunteers for testing bio-availability of Resveratrol containing supplement
- Laflavon group: Mixed age and gender group of healthy volunteers for testing bio-availability of Soy Isoflavones containing supplement

SUMMARY:
Cardiovascular disease (CVD) continues to rank high among the leading causes of morbidity and mortality in adults worldwide. While diet and increased physical activity constitute the primary preventive health approach, the role of plant-based bioactive compounds has attracted much attention due to their unique cardio-protective benefits. Several epidemiological studies suggest that dietary patterns characterized by relatively high intake of fruits and vegetables are significantly associated with reduced risks of coronary heart disease and stroke.

Dietary bioactive compounds are potent anti-oxidants and anti-inflammatory agents, thereby counteracting oxidative damage and inflammation, which underlie the pathogenesis of CVD.

However, this area is really lacking of a good set of chemistry, bioavailability and efficacy data that is vital for nutrition researchers and doctors to emphasize their role in the prevention and treatment of clinical outcomes at different stage of CVD, and dissemination of this information to the general public.

Cambridge Theranostics has focused its efforts on developing products that can prevent the damaging oxidation of lipoproteins that leads to heart attacks and stroke, and on understanding the cause of that damage.

Extensive literature shows that Lycopene, Resveratrol and Soy Isoflavones are key ingredients in diets that long been known to reduce the risk of heart attack and stroke. However, they are normally poorly absorbed (not 'bioavailable'). The investigators unique production process presents Lycopene, Soy Isoflavones and Resveratrol to the body in a form that it can easily absorb and use.

The aim of the current study is to perform and compare bioavailability and absorption of those three different dietary antioxidants and their combinations. The study is funded by Cambridge Theranostics and will be done on healthy volunteers of various ages with 30 people in each product group. It will be conducted on the primacies of Cambridge Theranostics in Babraham Research Campus. And managed by the team of experienced professionals employed by Cambridge Theranostics. The study will last about 12 months including recruitment process, screening process, periodical blood samples collection and examination and statistical analyses at the end.

DETAILED DESCRIPTION:
90 volunteers, who fulfill the inclusion criteria, do not meet any of the exclusion criteria, who have given written informed consent will be entered into the study. Lab assays and statistical analysis of the data will be performed on all plasma samples of those subjects who complete the study according to the study protocol or who partially complete the study with evaluable data. Subjects will be recruited from the subject pool of the CTL database.

The study will be performed as a daily for 8 weeks dose, open label, three arms study with 90 subjects.

The study will consist of three groups with one treatment period in each, with a wash-out period of 4 weeks prior the study.

All evaluable data are supposed to be used for the safety evaluation. The subjects will be taking products with a main meal daily. At certain time points (T0 - before study, T1 - 1 week of treatment, T2 - 2 weeks of treatment, T3 - 3 weeks of treatment, T4 - 4 weeks of treatment, T8 - 8 weeks of treatment) after an overnight fasting of about 11 hours the subjects will be invited to the lab for a blood sample collection. Blood samples for the analysis of serum concentrations of Lycopene, Resveatrol and Soy Isoflvones shall be drawn. Two aliquots of each sample will be prepared. One aliquot of each frozen serum sample will be shipped to analytical lab for bioanalysis of Lycopene, Resveatrol and Soy Isoflvones. Other aliquots will be retained at the CTL's lab. A total of 7 blood samples will be collected before and during product intake.

Analytical laboratory of Institute of Food Research, Norwich, will perform measurements of concentration of Lycopene, Resveatrol and Soy Isoflvones using a validated LC-MS/MS method. Calculations of the pharmacokinetic parameters and the assessment of bioavailability will be carried out for all products by CTL. The final report will include all aspects concerning the clinical part of the study, bioanalysis, statistics and discussion of obtained data as well as the legal and ethical requirements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, Caucasian male and female subjects 20 - 80.
* Female subjects of childbearing potential agree to undergo pregnancy tests and to use an appropriate method of contraception (i.e. oral contraceptive steroids, intrauterine device, barrier method).
* Findings within the range of clinical acceptability in medical history and physical examination, and laboratory results within the "normal ranges" for the relevant laboratory tests (unless the clinical investigator considers the deviation to be irrelevant for the purpose of the study).
* Normal vital signs, or abnormalities which the clinical investigator does not consider a disqualification for participation in the study.
* Willingness to undergo a pre-study physical examination and laboratory investigations.
* Ability to comprehend and willingness to sign both statements of informed consent (for screening and phase-related procedures).
* Non-smokers, mild to moderate smokers (≤ 10 cigarettes daily).

Exclusion Criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* History of or current compulsive alcohol abuse (> 10 drinks weekly), or regular exposure to other substances of abuse.
* Participation in another study with an experimental drug within 4 weeks before the first administration of study medication.
* A major illness during the 3 months before commencement of the screening period.
* History of hypersensitivity to the study product or any related products.
* History of bronchial asthma.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
* Donation or loss of blood equal to or exceeding 500 ml during the 8 weeks before the first administration of study medication or donation or loss blood from 250 to 500 ml in the 6 weeks before administration of study medication or donation or loss of blood up to 250 ml in the 4 weeks before administration of study medication.
* Resting heart rate of > 100 beats per minute or < 45 beats per minute during the screening period, either supine or standing.
* Positive testing for HIV and hepatitis B antigens.
* History of epilepsy
* Adverse events occurring in the pre-exposure phase, judged as "severe" by the principal investigator.
* Difficulty fasting or consuming the standard meals.
* Do not tolerate vein puncture.
* On a special diet within 4 weeks prior to drug administration (e. g. liquid, protein, raw food diet).
* Drug addiction requiring treatment in the past 12 months.
* Do not agree to fully participate in wash-out period and exclude from the diet the recommended food within 4 weeks before the study start and during the study.
* Tomato intolerants
* Milk intolerants

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Cambridgeshire
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
AUCt - Area under the serum concentration-time curve from the first time point [t=0] to the time point of the last measured concentration [t(last)] | 8 weeks
AUC∞ - Area under the serum concentration-time curve from the time point [t=0] to infinity [∞] | 8 weeks
Cmax - Maximum serum concentration | 8 weeks

SECONDARY OUTCOMES:
tmax - Time of maximum serum concentration | 8 weeks
t½ - Elimination half life
AUC(last)-∞ - Difference between AUC∞and AUCt expressed as percentage value
AUCt/AUC∞ - calculated as quotient of AUCt and AUC∞
f = Cmax/ AUCt (indication of rate of absorption)

CONTACTS AND LOCATIONS:
Locations (1):
- Babraham Research Campus, Cambridge, Cambridgeshire, United Kingdom